CLINICAL TRIAL: NCT01185704
Title: A Phase IIIb Randomized Open-label Study to Compare the Estradiol Level on the Releasing Day in Two Regimen of Cetrotide® 0.25 mg Used From Day 1 or From Day 7 of the Menstrual Cycle (Day 0 or Day 6 of Stimulation) in Polycystic Ovarian (PCO) Women in ART (IVF/ICSI).
Brief Title: Analysis of Two Therapeutic With Cetrotide® in Polycystic Ovarian (PCO) Women in Assisted Reproductive Technology (ART)
Acronym: ATTAC-PCO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.A.S, France (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR200088-501; 2007-007932-25 (EudraCT Number); INI 28091 (Other: Merck KGaA)
Record Dates: First submitted 2010-08-10; First posted 2010-08-20 (Estimated); Results first posted 2013-07-03 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Polycystic Ovarian Syndrome
Keywords: Cetrorelix acetate; follitropin alfa; human chorionic-gonadotropin alfa; follicular maturation; pregnancy; ovarian stimulation
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — cetrorelix; Chorionic Gonadotropin; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Day 1 protocol (Experimental)
  Interventions: Drug: Cetrorelix acetate; Drug: Recombinant Human Choriogonadotropin (r-hCG); Drug: Recombinant human follicle stimulating hormone (r-hFSH)
- Day 7 protocol (Experimental)
  Interventions: Drug: Cetrorelix acetate; Drug: Recombinant Human Choriogonadotropin (r-hCG); Drug: Recombinant human follicle stimulating hormone (r-hFSH)

INTERVENTIONS:
Drug: Cetrorelix acetate — Cetrotide® 0.25 mg will be administered subcutaneously once daily from Day 1 (Day 0 of stimulation period [S0]) until r-hCG day (at least 2 follicles >=17 mm)
  Other Names: Cetrotide®
  Arms: Day 1 protocol
Drug: Cetrorelix acetate — Cetrotide® 0.25 mg will be administered subcutaneously once daily from Day 7 (Day 6 of stimulation period [S6]) until r-hCG day (at least 2 follicles >=19 mm)
  Other Names: Cetrotide®
  Arms: Day 7 protocol
Drug: Recombinant Human Choriogonadotropin (r-hCG) — The r-hCG will be administered subcutaneously as a single dose of 250 microgram (mcg) on r-hCG day
  Other Names: Ovitrelle®
Drug: Recombinant human follicle stimulating hormone (r-hFSH) — Recombinant human follicle stimulating hormone (r-hFSH) will be administered subcutaneously at a dose between 75 and 187.5 international unit (IU) once daily from Day 2 (Day 1 of stimulation period [S1]) until r-hCG day

SUMMARY:
This is a randomized open-label study to compare between in-vitro fertilization/intracytoplasmic sperm injection (IVF/ICSI) outcomes of the two regimen of Cetrotide® (Cetrorelix acetate) which are 0.25 milligram (mg) used from Day 1 or Day 7 of the menstrual cycle (Day 0 or Day 6 of stimulation) in polycystic ovarian (PCO) women in assisted reproductive technology (ART).

DETAILED DESCRIPTION:
Polycystic ovarian syndrome population is an androgenic syndrome characterized by a wide spectrum of clinical manifestations such as obesity, hirsutism, insulin resistance, diabetes and presence of specific ultrasonic features.

Cetrotide®, cetrorelix acetate, is an antagonist of luteinizing-hormone-releasing hormone (LHRH). Cetrotide® is registered in 70 countries (including France) for the prevention of premature ovulation in subjects undergoing a controlled ovarian stimulation, followed by oocyte pick-up and ARTs. Ovitrelle®, active ingredient human chorionic-gonadotropin alfa, is administered to trigger final follicular maturation and luteinization after stimulation of follicular growth.

OBJECTIVES

Primary objective:

* To compare the hormonal level of plasmatic estradiol on the releasing day (day of r-hCG administration) induced by Cetrotide® 0.25 mg/day started on Day 1 (Group A: Day 1) or on Day 7 (Group B: Day 7) of the menstrual cycle (Day 0 (S0) or Day 6 (S6) of stimulation) in PCO subjects undergoing IVF/ICSI procedures.

Secondary objectives:

* To compare the hormonal changes during the stimulation induced by Cetrotide® in A and B Groups
* To assess by ultrasound scans (US) the follicular development induced by Cetrotide® in A and B Groups
* To assess biological and clinical outcomes induced by Cetrotide® in A and B Groups
* To monitor safety of Cetrotide in A and B Groups

The trial will be conducted on an outpatient basis. Once each subject has met all eligibility criteria, they will be randomly assigned in one of the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with PCO or Polycystic ovary syndrome (PCOS) according to the revised 2003 Rotterdam Consensus
* Female subjects suitable for IVF/ICSI, undergoing first or second attempt
* 18-35 years old, Body Mass Index (BMI) less than or equal to 32, non-smoking at least from Visit 0 (V0)
* Normal FSH value (less than 10 international unit per liter [IU/L]) on Day 3 of spontaneous cycle within 12 months prior to the trial
* Anti Mullerian Hormone (AMH) value (greater than 1.5 nanogram per milliliter [ng/mL]) of a spontaneous cycle within 12 months prior to the trial or at least at V0
* No history of active genito-urinary infection
* Normal thyroid function (or adequate substitution for at least 3 months)
* Negative cervical papanicolaou test within the last 12 months prior to study entry
* No gonadotropins, for at least one month prior to the trial
* No metformin therapy for at least one month prior to Visit 1 (V1)
* Subject who is able to participate in the trial and has provided written, informed consent.

Exclusion Criteria:

* Ongoing pregnancy, any pregnancy within 3 months prior to study entry, or any contraindication to pregnancy or carrying pregnancy to term
* Drilling 3 months prior to V0
* Uterine malformation, diethylstilbestrol syndrome, synechia
* Female subjects with World Health Organization (WHO) Type I or III anovulation
* Female subjects with hyperprolactinemia
* Female subjects with more than 2 recurrent miscarriages (early or late, and for any reasons)
* Known infection with Human Immunodeficiency Virus (HIV), Hepatitis B or C virus, for subject or partner
* Abnormal gynecological bleeding of undetermined origin
* History of major thromboembolic disease
* Endometriosis (Grade III or IV)
* Presence or history of malignant tumors and related treatment
* Known case of tumors of the hypothalamus or pituitary gland
* Clinically significant systemic disease or clinically significant abnormal hematology, chemistry, or urinalysis results at screening
* Known allergic reaction or hypersensitivity to Cetrotide® or Ovitrelle®
* Any active substance abuse or history of drug, medication or alcohol abuse in the past 5 years
* Participation in another clinical trial within 3 months prior to study entry.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2008-11; Primary Completion 2011-10 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Etienne VARLAN, Study Director — Merck Lipha Santé
Locations (1):
- Research Site, Toulouse, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Day 1 Protocol: Cetrotide® 0.25 milligram (mg) was administered subcutaneously once daily from Day 1 (Day 0 of stimulation period [S0]) along with Recombinant human follicle stimulating hormone (r-hFSH) at a dose between 75 and 187.5 international unit (IU) subcutaneously once daily from Day 2 (Day 1 of stimulation period [S1]) until recombinant human chorionic gonadotropin (r-hCG) administration day (at least 2 follicles greater than or equal to (>=) 17 millimeter [mm]). On r-hCG day, 250 microgram of r-hCG was administered once subcutaneously.
- Day 7 Protocol: Cetrotide® 0.25 mg was administered subcutaneously once daily from Day 7 (Day 6 of stimulation period [S6]) along with r-hFSH at a dose between 75 and 187.5 IU subcutaneously once daily from Day 2 (S1) until r-hCG administration day (at least 2 follicles >= 19 mm). On r-hCG day, 250 microgram of r-hCG was administered once subcutaneously.
Period: Overall Study
Arm/Group | Day 1 Protocol | Day 7 Protocol
Started | 68 | 68
Treated | 65 | 65
Completed | 55 | 60
Not Completed | 13 | 8
Not completed — Randomized but not treated | 3 | 3
Not completed — Lack of ovarian response | 5 | 1
Not completed — Ovarian hyperstimulation syndrome risk | 5 | 3
Not completed — Ectopic pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Day 1 Protocol | Day 7 Protocol | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (2.9) | 29.7 (3.3) | 29.7 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 65 | 130
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Estradiol (E2) Levels on r-hCG Day
Time Frame: r-hCG day (end of stimulation cycle [approximately 15 days])
Population: Intent to treat (ITT) population included all randomized participants who had received at least 1 dose of the study medication. N" (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | Day 1 Protocol | Day 7 Protocol
Number analyzed (Participants) | 58 | 62
picogram/milliliter (pg/mL) | 1668.86 (862.62) | 1672.80 (835.49)

2. Secondary Outcome: Serum Luteinizing Hormone (LH) and Follicle Stimulating Hormone (FSH) Levels
Time Frame: Day 1
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication. N" (number of participants analyzed) signifies those participants who were evaluable for this measure. Here "n" signifies those participants who were evaluated for specified category.
Measure: Mean (Standard Deviation); unit: International unit/liter (IU/L)
Arm/Group | Day 1 Protocol | Day 7 Protocol
Number analyzed (Participants) | 58 | 62
International unit/liter (IU/L)
  LH levels (n=58, 62) | 4.87 (4.62) | 6.84 (3.99)
  FSH levels (n=57, 59) | 4.98 (1.54) | 6.69 (10.29)

3. Secondary Outcome: Serum Estradiol (E2) Levels
Time Frame: Day 1
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Day 1 Protocol | Day 7 Protocol
Number analyzed (Participants) | 60 | 63
pg/mL | 30.42 (14.06) | 68.79 (116.09)

4. Secondary Outcome: Serum Progesterone (P4) Levels
Time Frame: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanomolar/liter (nmol/L)
Arm/Group | Day 1 Protocol | Day 7 Protocol
Number analyzed (Participants) | 59 | 62
nanomolar/liter (nmol/L) | 0.83 (0.72) | 0.97 (1.82)

5. Secondary Outcome: Anti Mullerian Hormone (AMH) Levels
Time Frame: Day 0
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Day 1 Protocol | Day 7 Protocol
Number analyzed (Participants) | 63 | 64
nanogram/milliliter (ng/mL) | 6.27 (4.40) | 7.18 (4.11)

6. Secondary Outcome: Number of Follicles Greater Than or Equal (>=) to 17 mm (For Day 1 Protocol) or 19 mm (For Day 7 Protocol) on r-hCG Day
Time Frame: r-hCG day (end of stimulation cycle [approximately 15 days])
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Day 1 Protocol | Day 7 Protocol
Number analyzed (Participants) | 58 | 61
follicles | 3.55 (2.20) | 2.49 (1.99)

7. Secondary Outcome: Number and Quality of Oocytes Retrieved
Description: Oocyte retrieval is a technique used in in-vitro fertilization (IVF) in order to remove oocytes from the ovary of the female participant, enabling fertilization outside the body. Oocytes were classified into 4 different categories based on their quality: mature, fractured, immature and inseminated oocytes.
Time Frame: Oocytes retrieval day (36 +/- 2 hours post r-hCG day [end of stimulation cycle {approximately 15 days}])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Day 1 Protocol | Day 7 Protocol
Number analyzed (Participants) | 65 | 65
oocytes
  Total number of oocytes | 7.48 (5.21) | 8.11 (5.55)
  Mature oocytes | 2.52 (4.07) | 3.72 (4.43)
  Fractured oocytes | 0.09 (0.34) | 0.11 (0.44)
  Immature oocytes | 0.98 (2.29) | 1.38 (2.55)
  Inseminated oocytes | 3.06 (4.14) | 4.52 (4.66)

8. Secondary Outcome: Total Dose of Recombinant Human Follicle Stimulating Hormone (r-hFSH)
Time Frame: Day 1 up to r-hCG day (end of stimulation cycle [approximately 15 days])
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: international unit (IU)
Arm/Group | Day 1 Protocol | Day 7 Protocol
Number analyzed (Participants) | 64 | 65
international unit (IU) | 1462.50 (537.85) | 1221.35 (478.31)

9. Secondary Outcome: Percentage of Fertilized Oocytes Retrieved
Description: Oocytes were fertilized using Intra-cytoplasmic Sperm Injection (ICSI) technique which is an IVF procedure in which a single sperm is injected directly into an egg under a microscope.
Time Frame: Oocytes retrieval day (36 +/- 2 hours post r-hCG day [end of stimulation cycle {approximately 15 days}])
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent fertilized oocytes
Arm/Group | Day 1 Protocol | Day 7 Protocol
Number analyzed (Participants) | 56 | 61
percent fertilized oocytes | 46.22 (30.66) | 46.86 (30.54)

10. Secondary Outcome: Number of Embryos
Description: Embryo is defined as the product of the zygote, two or three days after fertilization of the oocytes.
Time Frame: Day 2-3 post oocytes retrieval day (36 +/- 2 hours post r-hCG day [end of stimulation cycle {approximately 15 days}])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: embryos
Arm/Group | Day 1 Protocol | Day 7 Protocol
Number analyzed (Participants) | 65 | 65
embryos | 3.18 (3.18) | 3.60 (3.27)

11. Secondary Outcome: Number of Blastocysts
Description: Blastocyst is an embryo, five or six days after fertilization, with an inner cell mass, outer layer of trophectoderm and a fluid-filled blastocoele cavity.
Time Frame: Day 5-6 post oocytes retrieval day (36 +/- 2 hours post r-hCG day [end of stimulation cycle {approximately 15 days}])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: blastocysts
Arm/Group | Day 1 Protocol | Day 7 Protocol
Number analyzed (Participants) | 65 | 65
blastocysts | 0.26 (1.05) | 0.20 (0.90)

12. Secondary Outcome: Number of Transferred Embryos
Description: Embryo transfer is the procedure in which one or more embryos are placed in the uterus.
Time Frame: Day 2-3 post Oocytes retrieval day (36 +/- 2 hours post r-hCG day [end of stimulation cycle {approximately 15 days}])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: transferred embryos
Arm/Group | Day 1 Protocol | Day 7 Protocol
Number analyzed (Participants) | 65 | 65
transferred embryos | 0.95 (0.74) | 1.02 (0.74)

13. Secondary Outcome: Implantation Rate
Description: Implantation rate per reporting group was measured as the number of gestational sacs observed, divided by the number of embryos transferred multiplied by 100.
Time Frame: 5 weeks post oocytes retrieval day (36 +/- 2 hours post r-hCG day [end of stimulation cycle {approximately 15 days}])
Population: as for outcome 3
Measure: Number; unit: percent sacs per embryo
Arm/Group | Day 1 Protocol | Day 7 Protocol
Number analyzed (Participants) | 46 | 48
percent sacs per embryo | 36.90 | 32.25

14. Secondary Outcome: Percentage of Participants With Clinical Pregnancy
Description: Clinical pregnancy was defined as pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. It excludes ectopic pregnancy.
Time Frame: 10 weeks post r-hCG day (end of stimulation cycle [approximately 15 days])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Day 1 Protocol | Day 7 Protocol
Number analyzed (Participants) | 65 | 65
percentage of participants | 20 | 20

15. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered. A Serious Adverse Event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. To avoid the participant/event combination double-count AEs and SAEs are reported separately.
Time Frame: Day 1 up to end of study (15 days post last administration of study drug)
Measure: Number; unit: participants
Arm/Group | Day 1 Protocol | Day 7 Protocol
Number analyzed (Participants) | 65 | 65
participants
  AEs | 11 | 18
  SAEs | 2 | 4

ADVERSE EVENTS:
Time Frame: Day 1 up to end of study (15 days post last administration of study drug)
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Day 1 Protocol | Day 7 Protocol
Serious Adverse Events (participants affected / at risk) | 2/65 | 4/65
Other Adverse Events (participants affected / at risk) | 9/65 | 14/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Day 1 Protocol (N=65) | Day 7 Protocol (N=65)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Ovarian Hyperstimulation syndrome (Reproductive system and breast disorders) | 2 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Day 1 Protocol (N=65) | Day 7 Protocol (N=65)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Headache (Nervous system disorders) | 6 | 1
Injection site erythema (General disorders) | 1 | 1
Injection site irritation (General disorders) | 1 | 0
Injection site burning (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Ovarian Hyperstimulation syndrome (Reproductive system and breast disorders) | 0 | 6
Pelvic pain (Reproductive system and breast disorders) | 4 | 3
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Adnexa uterin pain (Reproductive system and breast disorders) | 1 | 0
Oestradiol increased (Investigations) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other